CLINICAL TRIAL: NCT04963972
Title: Impact of Digital and Behavioral Tele-Health Tapering Program for Perioperative Surgical Patients Exposed to Opioids
Brief Title: Digital and Behavioral Tele-Health Tapering Program for Lowering Dependence on Opioids in Patients Undergoing Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lucid Lane, Inc (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0769; NCI-2021-00053 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-02-24; First posted 2021-07-15 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Malignant Abdominal Neoplasm; Malignant Head and Neck Neoplasm; Malignant Solid Neoplasm; Malignant Thoracic Neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Behavior Therapy; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Lucid Lane) (Experimental): Patients participate in the Lucid Lane therapy program including working with a mental health therapist on mindfulness, CBT, group therapy, and mind-body therapies for 3-9 months or until the tapering off period is complete.
  Interventions: Behavioral: Behavioral Intervention; Other: Questionnaire Administration
- Arm II (standard of care) (Active Comparator): Patients receive standard of care post-surgical opioid education.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Participate in Lucid Lane therapy program
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (Lucid Lane)
Other: Best Practice — Receive standard of care opioid education
  Other Names: standard of care; standard therapy
  Arms: Arm II (standard of care)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the effect of behavioral health support including tele-health in helping surgical patients taper off of prescription opioid pain medications. "Tapering off" means taking dose amounts of medication that get smaller over time, so that less and less of the drug is used until it is not needed anymore. Researchers want to learn how these techniques may improve a patient's ability to lower or avoid dependence on opioid medications after surgery, and if behavioral therapies may improve quality of life, emotional well-being, and functional status around surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the impact of Lucid Lane's perioperative opioid tapering program utilizing daily behavioral health support (Health Insurance Portability and Accountability Act [HIPAA]-compliant sessions of cognitive behavioral therapy [CBT], mindfulness, 1:1 psychotherapy, group therapy, and 2-way texting and chat, all interactions with Lucid Lane licensed therapists), for patients who are on an opioid medication prior to surgery (tolerant), or naive and will be undergoing a surgery with curative intent post-surgery.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients participate in the Lucid Lane therapy program including working with a mental health therapist on mindfulness, CBT, group therapy, and mind-body therapies for 3-9 months or until the tapering off period is complete.

ARM II: Patients receive standard of care post-surgical opioid education.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Patients undergoing head and neck cancer surgery, open abdominal surgery, thoracic surgery
* Life-expectancy of 270 days or more
* Patients who will receive opioids as part of their treatment post-operatively
* Perioperative opioid use:

  * Naive Arm: No opioids 30 days prior to surgery
  * Tolerant Arm: Use of opioids on 2 or more days/week, for 1 or more months prior to surgery
* Patient is willing to use Lucid Lane program to provide behavioral health support perioperative period up to 9 months post-op for tolerant opioid users and 1 month for opioid naive users
* Patient is willing to discuss Lucid Lane progress with MD Anderson perioperative team and prescribing clinicians
* Patient is willing to sign a Lucid Lane Participant Agreement
* Patient is willing to sign an informed consent

Exclusion Criteria:

* Serious mental illnesses including schizophrenia-spectrum disorders, severe bipolar disorder, and severe major depression
* Active suicidal ideations
* Patients on methadone, naltrexone, or buprenorphine for treatment of opioid use disorder (i.e. for treatment of addiction, and not for treatment of pain)
* Patient unwilling to use or not possessing access to a device that allows for video visits (e.g. a smartphone, tablet, or computer)
* Patients who are on end-of-life care
* Insufficient ability to use English to participate in the consent process, the intervention or study assessments. The Lucid Lane therapists will be conducting therapy sessions in English, and the ability to understand English is required for the consent process. All questionnaires and surveys will be in English to ensure appropriate and comprehensive care for this patient population
* Insufficient ability to provide informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Percent tapered off of opioid in the telehealth group over time compared to usual care (opioid naive) | Up to 90 days
Percent tapered off of opioid in the telehealth group over time compared to usual care (opioid tolerant) | Up to 270 days

SECONDARY OUTCOMES:
Change in quality of life measures between telehealth group and usual care | Baseline up to 9 months
  Edmonton Symptom Assessment Scale (ESAS) Scale 0 symptom is absent up to Scale 10 symptom is worst possible severity, Brief Pain Inventory (BPI) Scale 0 no pain to Scale 10 pain at its worse, Patient Health Questionaire-9 (PHQ-9) Scale score totals: 1-4 minimal depression, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. EQ-5D-5L The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Change in emotional well-being (EWB) between telehealth group and usual care | Baseline up to 9 months
  Generalized Anxiety Disorder 7 item (GAD-7) scale Score totals of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. Further evaluation is recommended when the score is 10 or greater. Edmonton Symptom Assessment Scale (ESAS) Scale 0 symptom is absent up to Scale 10 symptom is worst possible severity. Patient Health Questionaire-9 (PHQ-9) 1-4 minimal depression, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. EQ-5D-5L The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Change in pain assessment between telehealth group and usual care | Baseline up to 9 months
  Edmonton Symptom Assessment Scale (ESAS) Scale 0 symptom is absent up to Scale 10 symptom is worst possible severity. Brief Pain Inventory (BPI) Scale 0 of no pain to scale 10 pain at its worse.
Change in satisfaction between telehealth group and usual care | Baseline up to 9 months
  Telehealth patient satisfaction survey. Scale range: Poor - Fair - Good - Excellent
Incidence of adverse events | Up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Koyyalagunta, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org